CLINICAL TRIAL: NCT01384201
Title: Evaluation of the Use of Confocal Endomicroscopy in Conjunction With Chromoendoscopy in the Detection of Gastric Preneoplastic Neoplasia and Neoplasia in a High-Risk Population (R-CE-GCEP)
Brief Title: Confocal Endomicroscopy Detection of Gastric Preneoplasia and Neoplasia
Acronym: R-CE-GCEP
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Associate Professor Yeoh Khay Guan, National University Health System, Singapore
Other Study IDs: NMRC/TCR/001/2007/CLE
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Gastric Intestinal Metaplasia
Keywords: intestinal metaplasia, gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — Biopsies from the stomach
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Confocal Laser Endomicroscopy: OGD by Confocal Endomicroscopy
- White light endoscopy: OGD by whitelight endoscopy

SUMMARY:
This is a prospective randomised study investigating the use of chromoendoscopy and confocal laser endomicroscopy for the detection of preneoplastic neoplasm in patients at high-risk of gastric cancer.

DETAILED DESCRIPTION:
This is a prospective randomised study investigating the use of chromoendoscopy and confocal laser endomicroscopy for the detection of preneoplastic neoplasm in patients at high-risk of gastric cancer. Patients are randomised to undergo upper endoscopy using either confocal laser endomicroscopy or standard whitelight endoscopy to investigate for gastric preneoplastic and neoplastic lesions.Results are compared to histopathologic diagnosis made on biopsies obtained during endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is Chinese
2. The subject is greater than 50 years of age
3. The subject satisfies one or more of the following criteria:

   * has (had) a history of dyspepsia of at least 4 weeks or more. Dyspeptic symptoms include bloating, epigastric discomfort and early satiety
   * has a family history of gastric cancer
   * has a medical condition for which an OGD is indicated.
4. The subject must have personally signed and dated the patient informed consent form indicating that he/she has been informed of all pertinent aspects of the study.
5. The subject must be willing and able to comply with scheduled visits and other study procedures

Exclusion Criteria:

1. The subject who has bleeding disorders, such as haemophilia, in whom biopsies are contraindicated.
2. The subject with liver cirrhosis.
3. The subject with previous total or partial gastrectomy.
4. The subject with severe co-morbid illness, such as end-stage renal failure (ESRF), congestive cardiac failure (CCF), severe osteoarthritis (OA) and rheumatoid arthritis (RA) requiring long term non-steroidal anti-inflammatory drug (NSAID) therapy.
5. The subject has other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may interfere with the interpretation of study results and in the judgment of the investigator would make the subject unsuitable for entry into the study.
6. The subject is currently on anti-coagulant therapy such as warfarin. Patients on aspirin, ticlopidine and clopidogrel must undergo a one-week washout period before enroling in the study.
7. The subject has a history of bronchial asthma, or a known allergy to fluorescein.
8. The subject is unwilling or unable to provide signed informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese, above 50 years old, at high risk of gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | On histopathologic diagnosis, usually 1-2 days after endoscopy
  The diagnostic yield, number of tissue biopsies per patient and percentage of missed lesions for CLE arm will be obtained by analyzing as though only targeted tissue biopsies are taken (CLE-TB), meaning that tissue biopsy is considered to have been performed only if the endoscopist gave the CLE diagnosis of GIM, dysplasia or malignancy. If the CLE diagnosis is normal, targeted tissue biopsy will be analyzed as not having been taken, and the corresponding histology for that site is for documenting any misdiagnosis by CLE in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Khay Guan Yeoh, MBBS; M Med, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore